CLINICAL TRIAL: NCT04738058
Title: Influence of Bovine Lactoferrin on Feeding Intolerance and Intestinal Permeability in Preterm Neonates: a Randomized Controlled Trial
Brief Title: Influence of Bovine Lactoferrin on Feeding Intolerance and Intestinal Permeability in Preterm Neonates
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Mansoura University Children Hospital (Other)
Responsible Party: Principal Investigator, Nermeen mohamed reda Mahmoud sameh Ellakany, Nermeen mohamed reda ellakany, Mansoura University Children Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MD.20.08.344
Record Dates: First submitted 2021-01-31; First posted 2021-02-04 (Actual); Last update posted 2021-02-04 (Actual); Status verified 2021-01

CONDITIONS: Feeding Intolerance in Preterm; Intestinal Permeability in Preterm
Keywords: Bovine lactoferrin; feeding intolerance; intestinal permeability; preterm
MeSH Terms: conditions — Premature Birth

STUDY DESIGN:
Intervention Model Description: Group A: preterm infants with feeding intolerance receive lactoferrin Group B: preterm infants with feeding intolerance receive placebo
Who Masked: Participant, Investigator
Masking Description: Closed sealed envelopes
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Preterm infants diagnosed as feeding intolerance will receive bovine lactoferrin (Experimental): they will receive bovine lactoferrin 100mg/day with feeding for 4 weeks or until discharge for preterm that was diagnosed as feeding intolerance
  Interventions: Drug: Bovine Lactoferrin Supplement
- Preterm infants diagnosed with feeding intolerance will receive placebo (Placebo Comparator): they will receive the placebo with feeding for 4 weeks or until discharge for preterm that was diagnosed as feeding intolerance
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: Bovine Lactoferrin Supplement — Bovine lactoferrin or placebo will be given to both arms with each feed for 30 days or till discharge from NICU the Lactoferrin dose 100mg/day Then determin is effect by serum zonulin level
  Other Names: Pravotin
  Arms: Preterm infants diagnosed as feeding intolerance will receive bovine lactoferrin
Drug: placebo — placebo
  Arms: Preterm infants diagnosed with feeding intolerance will receive placebo

SUMMARY:
Preterm infants are at increased risk of developing feeding intolerance due to functional immaturity of their gastrointestinal tract and may lead to discontinuation of enterak feeding.

Lactoferrin promotes the growth of probiotic bacteria, stimulates differntiation and proliferation of enterocytes and expression of intestinal digestive enzymes , lead to improvement of feeding intolerance.

So we hypothesized that supplementation of bovine lactoferrin would be benificial on feeding intolerance and decrease intestinal permeability in preterm infants with feeding intolerance.

DETAILED DESCRIPTION:
Preterm infants are at increased risk of developing feeding intolerance (FI) due to functional immaturity of their gastrointestinal tract. Feeding intolerance often leads to discontinuation of enteral feeds, delayed achievement of full enteral feeding, increased length of hospital stay, sub-optimal nutrition, postnatal growth restriction, prolonged parenteral feeding with an increased risk of nosocomial infections and poor neurodevelopmental outcome.1,2 Although there is no consensus on the definition of FI, a gastric residual volume of more than 50% of the previous feeding volume, gastric regurgitation, abdominal distension and/or emesis, are used as indicators for FI.1,3 Intestinal microflora plays an important role in the promotion and maintenance of intestinal functions such as mucosal trophism, gut barrier, sensori-motor function, hormone secretion, angiogenesis and immune defences.4 Many factors lead to unbalanced microflora colonization in the preterm infant as cesarean delivery, NICU stays, fasting and antibiotic use, leading to FI and necrotizing enterocolitis (NEC).5 Several strategies have been developed to improve the enteral feeding tolerance in preterm infants such as the implementation of standardized feeding protocols, the use of prokinetic agents and probiotics. The beneficial effect of probiotic supplementation on FI has been reported in several studies.6,7 Multiple mechanism of action has been proposed, including strengthening the intestinal mucosal barrier function, thereby inhibiting bacterial translocation, regulation of bacterial colonization, modulation of intestinal inflammation.8 Although probiotics may be a promising approach for the prevention of FI and NEC in preterm infants, several issues exist regarding strain specificity, schedule of supplementation, and long-term adverse effects.9 Lactoferrin (LF), a member of the transferrin family of iron-binding glycoproteins, is present in high amounts in colostrum and maternal milk.

Lactoferrin is almost completely absent from processed formulae. Lactoferrin is the major factor responsible for the protective effects of breast milk-decreased rates of infection and NEC, improved neurodevelopment and better immune responses due to its antimicrobial, anti-oxidant, anti-inflammatory and immunomodulatory properties.10 Lactoferrin stimulates gastrointestinal cell proliferation and differentiation via extracellular signal-regulated kinase, limits IL-8 secretion, prevents NF-kB and hypoxia-inducible factor-1a activation, suggesting strong anti-inflammatory effects.11 Lactoferrin also promotes the growth of probiotic bacteria, stimulates differentiation and proliferation of enterocytes and expression of intestinal digestive enzymes.12 Its bifidogenic activity in the gut may improve tolerance to feeds.13 Very preterm infants receive little or no milk during early neonatal period and have low intake of LF.14 Because human LF is expensive, bovine lactoferrin has been considered as an alternate supplement to correct this deficiency, as it is about 70% homologous with human LF but has higher antimicrobial activity.15 Bovine LF has no known toxicity and is registered as GRAS (Generally Recognised As Safe) by the US Food and Drug Administration.16 A systematic review including 6 RCTs involving almost 1100 preterm infants concluded that there is an evidence of low quality suggesting that LF supplementation to enteral feeds with or without probiotics decreases late-onset sepsis and NEC stage II or III in preterm infants without adverse effects.17 A more recent systematic review, included 9 trials that enrolled 1834 preterm infants indicated that LF supplementation in preterm neonates is safe without obvious adverse effects, could significantly reduce the incidence of NEC, and hospital-acquired infection. Moreover, LF could reduce the time to achieve full enteral feeding (the mean difference for days to achieve full enteral feeding in preterm infants was -2.19 days) and duration of hospitalization of preterm infants.18 A large RCT "The ELFIN Trial", included 2203 infants, has demonstrated that enteral LF supplementation (150 mg/kg per day until 34 weeks' postmenstrual age) does not reduce the risk of late-onset infection, other morbidity, or mortality in very preterm infants. However, this study did not rule out important potential benefits, particularly for infants who receive formula for over half of days of enteral feeds.19 The intestinal barrier provides highly selective protection of the human body against the environment. It has several facets, which include: intestinal microbiota; a protective mucus layer; intestinal epithelium cells with tight junctions (TJ); and cells of the immune system and enteric nervous system.20 Intestinal barrier maturation in preterm infants is gestational age and postnatal age-dependent and is influenced by feeding type and antibiotic exposure.21 Zonulin (ZO), is an established marker of intestinal permeability. Zonulin is one of the proteins that regulate the function of TJ between intestinal epithelial cells, which determines paracellular transport in the gut. It is one of the main factors securing the action of the "gate of the gut" mechanism by reversibly influencing TJ's tightness. Zonulin increase and disruption of TJ has been demonstrated in an animal model of NEC with intestinal TJ destruction proven by immune histochemical evaluation.22 Zonulin increases in newborns presenting symptoms of infection and/ or inflammation of the gut or being at risk of intestinal pathology.23 We hypothesized that supplementation of bovine LF would have beneficial effects on feeding tolerance and decrease intestinal permeability in preterm infants with FI.

ELIGIBILITY:
Inclusion Criteria:

* preterm infants delivered at gestational age 26 to 34 weeks admitted to NICU OF mansoura university children hospital Diagnosed as feeding intolerance defined as gastric volume residual of more than 50% of the previous feeding volume, gastric regurgitation, abdominal distention and or emesis Receive premature cow's protein based formula enteral feeding

Exclusion Criteria:

Major congenital malformations Anatomical gastrointestinal anomalies Birth asphyxia Presence of NEC Neonate receiving Expressed breast milk Infant with history of cow's milk allergy

-

Ages: 26 Weeks to 34 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Estimated)
Dates: Start 2020-12-15 (Actual); Primary Completion 2021-12 (Estimated); Study Completion 2022-06 (Estimated)

PRIMARY OUTCOMES:
Duration required by the infant to achieve full enteral feeding | 4 weeks or till discharge from NICU, whichever came first
  Full enteral feed reached when infant tolerated 150ml/kg/day
Serum zonulin concentrations at day 7 and 4 weeks after enrollment or discharge | 4 weeks or till discharge from NICU, whichever came first
  serum zonulin is an indicator for intestinal permeability

SECONDARY OUTCOMES:
Number of episodes of gastric residual more than 50% of the previous feed | 4 weeks or till discharge from NICU, whichever came first
  Number of episodes of gastric residual more than 50% of the previous feed
Weight gain | 4 weeks or till discharge from NICU, whichever came first
  weight gain during admission
Late onset sepsis | 4 weeks or till discharge from NICU, whichever came first
  by sighs and Lab. investigation of sepsis
Total numbers of days of antimicrobial administration | 4 weeks or till discharge from NICU, whichever came first
  Total numbers of days of antimicrobial administration
Duration of parenteral nutrition | 4 weeks or till discharge from NICU, whichever came first
  during NICU stay
Necrotizing enterocolitis | 4 weeks or till discharge from NICU, whichever came first
  Bell stage 2 or 3
Duration of hospital stay | 4 weeks or till discharge from NICU, whichever came first
  Duration of hospital stay
Iron status after 4 week of enrollment | 4 weeks or till discharge from NICU, whichever came first
  serum iron , serum ferritin, TIBC
Side effect from the drug | 4 weeks or till discharge from NICU, whichever came first
  vomiting , rash

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed M Hassan, Professor, Study Director — Mansoura University Children Hospital; Hesham S Abd El Hady, Study Director — Mansoura University Children Hospital
Locations (1):
- Mansoura University Children Hospital, Al Mansurah, Egypt

REFERENCES:
- [Derived] Ellakkany N, Abdel-Hady H, Eita AM, Mosaad YM, Megahed A. Influence of bovine lactoferrin on feeding intolerance and intestinal permeability in preterm infants: a randomized controlled trial. Eur J Pediatr. 2024 Nov 20;184(1):30. doi: 10.1007/s00431-024-05861-4. PMID 39565449
- See also: Prophylactic lactoferrin for preventing late-onset sepsis and necrotizing enterocolitis in preterm infants — https://www.ncbi.nlm.nih.gov/pmc/articles/PMC6392939/